CLINICAL TRIAL: NCT02788877
Title: Single Arm, Single Dose Clinical Study to Investigate Efficacy of Treat-and-Extend Regimen of Intravitreal Aflibercept Injection in Diabetic Macular Edema
Brief Title: Treat-and-extend Regimen of Aflibercept in Diabetic Macular Edema (VIBIM Study)
Acronym: VIBIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Ji Eun Lee, Professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160043
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Macular Edema, Diabetic
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treat-and-extend (Experimental): Aflibercept 2mg is injected into the vitreous cavity. An injection is given every 4 weeks five times and then the Treat-and-Extend process begins. If 1mm central subfield macular thickness (CSMT) improved (10% or more reduction) compared to the previous visit, the next treatment will be performed at the same interval. If CSMT is maintained (less than 10% changes), the next interval will be extended by two weeks (up to 12 weeks). If CSMT is worsened (10% or more increase), the next interval will be shortened by two weeks (minimum 4 weeks). If CSMT is stable two times at 12 weeks-interval, the injection will be deferred, and the next visit will be 8 weeks later. These process will be continued for 2 years.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — Aflibercept 2mg is injected into the vitreous cavity through the pars plana using 30 gauge needle-attached syringe.
  Other Names: Eylea, VEGF Trap-Eye

SUMMARY:
Efficacy of Treat-and-extend regimen (TER) using aflibercept in diabetic macular edema (DME) will be evaluated.

DETAILED DESCRIPTION:
Efficacy of aflibercept for diabetic macular edema was demonstrated in the phase III, VIVID and VISTA studies. In these studies, aflibercept was injected using the fixed dosing regimen that an intravitreal injection was performed 5 times every 4 weeks and then every 8 weeks. Although the efficacy was comparable to that of ranibizumab injected every 4 weeks, continuous visits and treatments account for quite a burden. TER is regarded as a alternative regimen that may reduce visit and treatment numbers for age-related macular degeneration. TER is a variable dosing regimen that an injection interval is adjusted based on the treatment response. The aim of this study is to evaluate efficacy of TER using aflibercept for DME, by assessing changes of visual acuity at 104 weeks compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Type I or II diabetes older than 18 years old
2. Patients with DME secondary to diabetes mellitus involving the center of the macula (defined as CSMT >= 300μm measured using OCT) in the study eye.
3. Decreased visual acuity to 20/40 - 20/300 to be primarily the results of DME in the study eye.
4. Willing and able to comply with clinic visits and study-related procedures, and provide a signed informed consent form.

Exclusion Criteria:

1. History of vitreoretinal surgery including scleral buckling in the study eye.
2. Laser photocoagulation (panretinal or macular) in the study eye within 90 days of day 1.
3. More than two previous macular laser treatments in the study eye.
4. Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of day 1.
5. Previous treatment with anti-angiogenic drugs in the study eye within 90 days of day 1.
6. Active proliferative diabetic retinopathy in the study eye.
7. History of idiopathic or autoimmune uveitis in the study eye.
8. Cataract surgery within 90 days before day 1 in the study eye.
9. Aphakia in the study eye.
10. Yttrium-aluminium-garnet capsulotomy in the study eye within 30 days before day 1.
11. Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or on OCT that is thought to affect central vision.
12. Current iris neovascularization, vitreous hemorrhage, or tractional retinal detachment in the study eye.
13. Structural damage to the center of the macula in the study eye that is likely to preclude improvement in best-corrected visual acuity (BCVA) following the resolution of macular edema including atrophy of the retinal pigment epithelium, subretinal fibrosis or scar, significant macular ischemia or organized hard exudates.
14. Evidence of infection including infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye.
15. Uncontrolled glaucoma in the study eye (>25mmHg) or filtration surgery and/or valve surgery for glaucoma in the past on the study eye.
16. Myopia of a spherical equivalent prior to any possible refractive or cataract surgery of ≥ -8 diopters.
17. Concurrent disease in the study eye, other than DME, that could compromise VA, require medical or surgical intervention during the study period, or could confound interpretation of the results (including retinal vascular occlusion retinal detachment, macular hole, or choroidal neovascularization of any cause).
18. Ocular media of insufficient quality to obtain fundus and OCT images.
19. Current treatment for a serious systemic infection.
20. Administration of systemic anti-angiogenic agents within 180 days before day 1.
21. Uncontrolled diabetes mellitus in the opinion of the investigator (VISTA) or as defined by hemoglobin A1c >12%.
22. Uncontrolled blood pressure (defined as systolic >160 mmHg or diastolic > 95 mmHg while patient is sitting).
23. History of either cerebral vascular accident and/or myocardial infarction within 180 days prior to day 1.
24. Renal failure requiring dialysis or renal transplant.
25. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, might affect interpretation of the results of the study, or renders the patient at high risk for treatment complications.
26. Pregnant or breast-feeding women.
27. Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study.
28. Allergy to fluorescein.
29. Patients with hypersensitivity to study drug or excipients.
30. Participation in an investigational study within 30 days prior to screening visit that involved treatment with any drug (excluding vitamins and minerals) or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-04-10 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in visual acuity from baseline to 104 weeks | baseline and 104 weeks
  Visual acuity is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Visual acuity of 85 letters is equivalent to 20/20. Higher scores represents better functioning.

SECONDARY OUTCOMES:
Changes in visual acuity from baseline to 52 weeks | baseline and 52 weeks
  Visual acuity is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Visual acuity of 85 letters is equivalent to 20/20. Higher scores represents better functioning.
Changes in CSMT from baseline to 104 weeks | baseline and 104 weeks
  CSMT is central 1mm thickness of the macula measured using spectral-domain optical coherence tomography (OCT). Normal thickness is around 250μm. Increased CSMT is regarded as presence of macular edema.
Number of injections for 52 and 104 weeks | 52 and 104 weeks
  How many injections are performed from baseline to 52 and 104 weeks.
Injection interval | 52 and 104 weeks.
  The interval is calculated for the next visit based on the treatment response. The range is between 4 and 12 weeks.
Percentage of patients with injection interval of 12 weeks or more | 104 weeks.
  Patients whose injection interval is extended to 12 weeks more include the patients that the next visit was calculated as 12 weeks and those that the injection was deferred in the previous visit.
Percentage of patients that visual acuity increased 15 letters or more | baseline, 52 and 104 weeks.
  Visual acuity was assessed using ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. Percentage of patients whose visual acuity increased 15 letters or more compared to baseline will be calculated.
Percentage of Patients With Visual Acuity >=20/40 | 52 and 104 weeks
  Visual acuity was assessed using ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. Percentage of patients with visual acuity 70 ETDRS letters (equivalent to 20/40) or better was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Pil Shin, MD, PhD, Study Director — Kyungbuk National University Hospital
Locations (8):
- South Korea (8):
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Haeundae Paik Hospital, Busan
  - Busan Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Gupta OP, Shienbaum G, Patel AH, Fecarotta C, Kaiser RS, Regillo CD. A treat and extend regimen using ranibizumab for neovascular age-related macular degeneration clinical and economic impact. Ophthalmology. 2010 Nov;117(11):2134-40. doi: 10.1016/j.ophtha.2010.02.032. Epub 2010 Jul 1. PMID 20591490
- [Background] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915